CLINICAL TRIAL: NCT03470584
Title: Vegetarian Diet and Chronic Degenerative Diseases in the Tzu Chi Health Study (TCHS) and the Tzu Chi Vegetarian Study (TCVS)
Brief Title: Vegetarian Diet and Chronic Degenerative Diseases
Status: Completed | Type: Observational
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TCHS-02
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2018-03

CONDITIONS: Dementia; Depression; Cardiovascular Diseases; Stroke; Gout; Cataract; Gallstone; Urinary Tract Infections
Keywords: Diet, vegetarian; Dementia; Depression; Cardiovascular Diseases; Stroke; Gout; Cataract; Gallstone; Urinary Tract Infections
MeSH Terms: conditions — Dementia; Depression; Cardiovascular Diseases; Stroke; Gout; Cataract; Gallstones; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for 3500 participants from the Tzu Chi Health Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tzu Chi Vegetarian Study: 12062 Tzu Chi volunteers of the Buddhist Tzu Chi Foundation recruited throughout communities in Taiwan in the year 2005. All participants filled out a self-administered questionnaire on basic information, medical history, lifestyle, and diet. Diet exposure: 1/3 vegetarians, 2/3 nonvegetarians.
  Interventions: Other: Diet Exposure
- Tzu Chi Health Study: 6002 participants who came for health examination at the Dalin Tzu Chi Hospital between the years 2007 to 2009. 77% were Tzu Chi volunteers. All participants were interviewed on a structured questionnaire including basic information, medical history, lifestyle, and diet, and received a comprehensive health examination. Diet exposure: 1/3 vegetarians, 2/3 nonvegetarians.
  Interventions: Other: Diet Exposure

INTERVENTIONS:
Other: Diet Exposure — Vegetarian diet vs nonvegetarian diet

SUMMARY:
To investigate the prospective association between a vegetarian diet and chronic degenerative diseases in two cohorts of Taiwanese Buddhists

DETAILED DESCRIPTION:
The Tzu Chi Vegetarian Study (TCVS) recruited 12062 community volunteers of the Buddhists Tzu Chi Foundation throughout Taiwan in the year 2005. All participants completed a self-administered questionnaire on basic information, medical history, lifestyle, and diet.

The Tzu Chi Health Study (TCHS) recruited 6002 participants who came to the Buddhist Tzu Chi Dalin General Hospital for health examination. All participants were interviewed on basic information, medical history, lifestyle, and diet. Biochemical and anthropometric data was collected through a health examination:

Biochemical variables: CBC, fasting glucose, lipid profile (TCH, LDL, HDL, TG), BUN, Cr, ALT, AST, and UA. In addition, homocysteine, serum vitamin B12, folate, and C-reactive protein (CRP) are available for 1500 subjects.

Blood: Extra blood samples have been obtained and stored for 3500 subjects and will be available for future investigation.

Anthropometric variables: body weight, height, waist circumference, % body fat (with BIA), blood pressure, pulse wave velocity, bone mineral density through DXA (at spine for female and hip for male), lung function test (spirometric), abdominal sonography, colonoscopy, esophageal-gastro-duodenal-scopy, chest X-ray, KUB.

Follow-up: Individual baseline data were linked to the National Health Insurance Database and the National Death Registry to ascertain disease outcomes at the Health and Welfare Data Science Center.

ELIGIBILITY:
Inclusion Criteria:

* Participants who consent to be followed.

Exclusion Criteria:

* Participants with inaccurate ID which make linkage to NHIRD impossible.
* Participants already with study outcome (disease) prior to enrollment in the study.
* Participants with missing covariates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the Tzu Chi Vegetarian Study were all certified volunteers of the Buddhist Tzu Chi Foundation. Participants of the Tzu Chi Health Study were the ones who came to the Dalin Tzu Chi Hospital for health examination and agree to join the cohort study (77% were certified Tzu Chi volunteers). About 1/3 of both cohorts were vegetarians at enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 18064 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2005-12-30 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Gout | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of gout are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of gout are identified using ICD-9 code: 274.
Stroke | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of stroke are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of stroke are identified using ICD-9 code: 430-438, where hemorrhagic stroke is defined by ICD9 430-432 and ischemic stroke is defined by ICD9 433-434.
Cataract | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of cataract are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of cataract are identified using ICD-9 code: 366.
Gallstone disease | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of gallstone disease are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of gallstone diseases are identified using ICD-9 code: 574.
Dementia and mild cognitive impairment | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of dementia are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of dementia and mild cognitive impairment are identified using ICD-9 code: 290.0, 290.1,290.4, 331.0, 331.1, 331.82, 331.83.
Depression | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of depression are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of depression and are identified using ICD-9 code: 296.2, 296.3, 300.4 and 311.
Urinary tract infections (UTI) | From enrollment to time of disease occurrence, death of any cause, or end of study period (December 31st 2014).
  Incidence of UTI are ascertained by linking individual participants' baseline data to the the National Health Insurance Database. Cases of UTI are identified using ICD-9 code: 599.0, 595, 590.
Medical expenditures | From enrollment to December 31st 2014.
  Actual medical expenditure associated with different dietary patterns are analyzed. Medical expenditures are obtained and computed from the National Health Insurance Database claim data for outpatient treatment, inpatient treatment, and dental treatment. This also includes costs associated with laboratory work and medication prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Lon Lin, MD, Study Chair — Dalin Tzu Chi General Hospital
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The disease outcome data from the National Health Insurance Database belongs to the Ministry of Health in Taiwan. Access to these data requires permission and formal application to the Health and Welfare Data Science Center, Ministry of Health in Taiwan. This is regulated by local law and regulation to protect individual personal information. Our research team does not have the right to release any data other than summarized results in the forms of peer-reviewed publications, for noncommercial purposes.

REFERENCES:
- [Background] Chiu THT, Liu CH, Chang CC, Lin MN, Lin CL. Vegetarian diet and risk of gout in two separate prospective cohort studies. Clin Nutr. 2020 Mar;39(3):837-844. doi: 10.1016/j.clnu.2019.03.016. Epub 2019 Mar 27. PMID 30955983
- [Background] Chiu THT, Chang HR, Wang LY, Chang CC, Lin MN, Lin CL. Vegetarian diet and incidence of total, ischemic, and hemorrhagic stroke in 2 cohorts in Taiwan. Neurology. 2020 Mar 17;94(11):e1112-e1121. doi: 10.1212/WNL.0000000000009093. Epub 2020 Feb 26. PMID 32102976
- [Background] Chiu THT, Chang CC, Lin CL, Lin MN. A Vegetarian Diet Is Associated with a Lower Risk of Cataract, Particularly Among Individuals with Overweight: A Prospective Study. J Acad Nutr Diet. 2021 Apr;121(4):669-677.e1. doi: 10.1016/j.jand.2020.11.003. Epub 2020 Dec 11. PMID 33309591
- [Background] Chang CM, Chiu THT, Chang CC, Lin MN, Lin CL. Plant-Based Diet, Cholesterol, and Risk of Gallstone Disease: A Prospective Study. Nutrients. 2019 Feb 4;11(2):335. doi: 10.3390/nu11020335. PMID 30720747
- [Background] Lin CL, Wang JH, Chang CC, Chiu THT, Lin MN. Vegetarian Diets and Medical Expenditure in Taiwan-A Matched Cohort Study. Nutrients. 2019 Nov 6;11(11):2688. doi: 10.3390/nu11112688. PMID 31698872
- [Background] Chen YC, Chang CC, Chiu THT, Lin MN, Lin CL. The risk of urinary tract infection in vegetarians and non-vegetarians: a prospective study. Sci Rep. 2020 Jan 30;10(1):906. doi: 10.1038/s41598-020-58006-6. PMID 32001729